CLINICAL TRIAL: NCT03885024
Title: The Peer-Based Retention of People Who Use Drugs in Rural Research
Acronym: PROUD-R2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Kentucky (Other); Ohio State University (Other); Emory University (Other); University of North Carolina (Other)
Responsible Party: Principal Investigator, P. Todd Korthuis, MD, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PROUD-R2
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Drug Use; Peer Influence

STUDY DESIGN:
Intervention Model Description: This study proposes a two-arm, individual-level randomized trial in which those in the intervention condition refer a "study buddy" peer who will be trained to help retain the index participant in their follow-up visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retention Video (Active Comparator): Participants the peer-driven retention arm will receive video-based and in-person training from Retention Specialists on how to encourage study retention. Participants will watch a 7 minute video that standardizes retention messages. A brief face-to-face conversation with the Retention Specialist follows the video viewing to answer questions and reinforce video messages. At the end of the training, participants receive information about their recruit(s) who consented to release their information to their recruiters. Peers remind their enrolled "study buddy" to attend their scheduled follow up assessments. Participants meet with a study Retention Specialist by phone or in person, at 3 and 9 months after enrollment to answer questions about peer retention strategies and remind participants of their peers' contact information and follow-up schedules.
  Interventions: Other: Retention Video
- Standard Retention Strategy (No Intervention): Control arm: At NROI enrollment, all participants provide detailed information to assist with retention and/or contact for future research, and contact information for up to three people who should know how to reach the participant if contact information changes. Participants randomized to receive the standard retention strategy are contacted at the mid-point of each follow-up interval (i.e., at 3-month post enrollment and 9-months post-enrollment) to update locator information and remind them about their follow-up appointment date. Study associates contact the participant using their contact information and, if not successful, will try to reach one of their contacts in the locator form.

INTERVENTIONS:
Other: Retention Video — Participants assigned to the retention training arm will watch a brief training video that will include information on how to retain peers in clinical trials.
  Arms: Retention Video

SUMMARY:
The purpose of this study is to, through several aims, test the effectiveness of peer-driven intervention and inform methods to optimize engagement in research in people who use drugs (PWUD) in rural America.

DETAILED DESCRIPTION:
This study builds on the National Rural Opioids Initiative (NROI), a multi-state consortium studying access to care, overdose, and infectious consequences of opioid use disorder (OUD) in Rural America. It includes counties in rural Oregon and Appalachian Kentucky and Ohio with high rates of drug overdose.

Aim 1: Conduct a randomized trial to evaluate the effectiveness of a peer-driven study retention intervention for retaining PWUD in Kentucky, Ohio, and Oregon Rural Opioid Initiative sites.

Aim 2: Elicit preferences of PWUD in the Kentucky, Ohio, and Oregon Rural Opioid Initiative sites Aim 2a: Administer baseline survey of discrete choice experiment preferences for participating in clinical trials of potential medical innovations (e.g. new treatments for OUD, HIV, and HCV vaccination). Aim 2a will be accomplished as part of the NROI studies. The data will then be merged for PROUD-R² analyses.

Aim 2b: Compare participant survey preferences regarding willingness to participate in clinical trials at baseline, 6, and 12 months.

Aim 3: Explore participant perceptions of clinical research participation and retention among PWUD in rural America.

ELIGIBILITY:
Inclusion Criteria:

NROI eligibility criteria: Participants are eligible to enroll in the NROI if they 1) live in the study area, 2) have recently injected drugs or report opioid use to get high without injection, and 3) are age 18 or older.

NROI participants enrolled after April 2019 are eligible to participate in the PROUD R2 study.

Participants enrolling as study buddies will be eligible if they 1) live in the study area, 2) are age 18 or older; they do not need to have recent or past substance use to qualify.

No eligible participants are excluded.

Exclusion Criteria:

Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
12 Month Retention Rate | 12 months
  Participants receiving the peer retention intervention will have 20% higher retention at 12 months (primary outcome) than those receiving the standard retention approach, alone.

SECONDARY OUTCOMES:
6 Month Retention Rate | 6 months
  Participants receiving the peer retention intervention will have higher retention at 6 months (secondary outcome) compared with those receiving the standard retention approach, alone.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Korthuis, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young AM, Lancaster KE, Bielavitz S, Elman MR, Cook RR, Leichtling G, Freeman E, Estadt AT, Brown M, Alexander R, Barrie C, Conn K, Elzaghal R, Maybrier L, McDowell R, Neal C, Lapidus J, Waddell EN, Korthuis PT. Peer-based Retention Of people who Use Drugs in Rural Research (PROUD-R2): a multisite, randomised, 12-month trial to compare efficacy of standard versus peer-based approaches to retain rural people who use drugs in research. BMJ Open. 2022 Jun 15;12(6):e064400. doi: 10.1136/bmjopen-2022-064400. PMID 35705346